CLINICAL TRIAL: NCT01005251
Title: Investigate the Effect of Different Doses of Lesogaberan (AZD3355) as add-on to PPI in GERD Patients With Partial Response to PPI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9120C00019
Record Dates: First submitted 2009-10-27; First posted 2009-10-30 (Estimated); Results first posted 2011-04-25 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-03

CONDITIONS: Gastroesophageal Reflux Disease; Heartburn; Regurgitation
Keywords: GERD treatment; Acid and non-acid Reflux; Heartburn; Regurgitation; Add-on treatment to PPI
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — lesogaberan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 60 mg (Experimental): PPI+lesogaberan (AZD3355) 60 mg bid
  Interventions: Drug: lesogaberan (AZD3355)
- 120 mg (Experimental): PPI+lesogaberan (AZD3355) 120 mg bid
  Interventions: Drug: lesogaberan (AZD3355)
- 180 mg (Experimental): PPI+lesogaberan (AZD3355) 180 mg bid
  Interventions: Drug: lesogaberan (AZD3355)
- 240 mg (Experimental): PPI+lesogaberan (AZD3355) 240 mg bid
  Interventions: Drug: lesogaberan (AZD3355)
- Placebo (Placebo Comparator): PPI+ Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lesogaberan (AZD3355) — 60 mg, oral, capsules, bid for 4 w
  Arms: 60 mg
Drug: lesogaberan (AZD3355) — 120 mg, oral, capsules, bid for 4 w
  Arms: 120 mg
Drug: lesogaberan (AZD3355) — 180 mg, oral, capsules, bid for 4 w
  Arms: 180 mg
Drug: lesogaberan (AZD3355) — 240 mg, oral, capsules, bid for 4 w
  Arms: 240 mg
Drug: Placebo — oral,capsules, bid for 4 w
  Arms: Placebo

SUMMARY:
This study is being carried out to see whether AZD3355 is an effective treatment as an add-on to PPI therapy in patients with Gastroesophageal Reflux Disease (GERD) with a partial response to PPI and to compare this with Proton Pump Inhibitor (PPI) treatment alone. Another goal of the study is to examine which of the investigated doses of AZD3355 is optimal for treatment of these patients. This study will also measure levels of drug in the blood and see how well it is tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Have at least 6 months history of GERD
* Continuously treated during the last 4 weeks before enrolment with daily optimized unchanged PPI therapy for any GERD indication

Exclusion Criteria:

* Patients that have not experienced any GERD symptom improvement at all during PPI treatment
* Prior surgery of the upper gastrointestinal tract.
* Subject who have any of the following conditions or diseases: Heart disease, Angina, Seizure disorders such as epilepsy, Congestive Heart Failure (CHF), Liver disease such as Cirrhosis or Hepatitis, Kidney disease, Lung disease or lung cancer, Cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 661 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Silberg, MD, Study Director — AstraZeneca; Nicholas Shaheen, MD, MPH, Principal Investigator — UNC Hospitals, 4141Chapel Hill, NC 27599 USA
Locations (1):
- Research Site, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Shaheen NJ, Denison H, Bjorck K, Silberg DG. Esophageal mucosal breaks in gastroesophageal reflux disease partially responsive to proton pump inhibitor therapy. Am J Gastroenterol. 2013 Apr;108(4):529-34. doi: 10.1038/ajg.2012.447. Epub 2013 Jan 15. PMID 23318482
- [Derived] Shaheen NJ, Denison H, Bjorck K, Karlsson M, Silberg DG. Efficacy and safety of lesogaberan in gastro-oesophageal reflux disease: a randomised controlled trial. Gut. 2013 Sep;62(9):1248-55. doi: 10.1136/gutjnl-2012-302737. Epub 2012 Jun 23. PMID 22730470

RESULTS

PARTICIPANT FLOW:
Groups:
- AZD3355 60 mg: PPI+AZD3355 60 mg twice daily (bid)
- AZD3355 120 mg: PPI+AZD3355 120 mg twice daily (bid)
- AZD3355 180 mg: PPI+AZD3355 180 mg twice daily (bid)
- AZD3355 240 mg: PPI+AZD3355 240 mg twice daily (bid)
- Placebo: PPI+Placebo
Period: Overall Study
Arm/Group | AZD3355 60 mg | AZD3355 120 mg | AZD3355 180 mg | AZD3355 240 mg | Placebo
Started | 134 | 125 | 136 | 126 | 140
Completed | 121 | 109 | 114 | 114 | 122
Not Completed | 13 | 16 | 22 | 12 | 18
Not completed — Withdrawal by Subject | 2 | 5 | 3 | 4 | 9
Not completed — Eligibility criteria not fulfilled | 4 | 0 | 4 | 1 | 0
Not completed — Adverse Event | 2 | 6 | 8 | 5 | 4
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 2
Not completed — Developed study-specific withdrawal crit | 2 | 0 | 3 | 0 | 1
Not completed — Lost to Follow-up | 1 | 4 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2
Not completed — Patient moved | 1 | 0 | 0 | 0 | 0
Not completed — Wrong drug dispensed | 0 | 1 | 0 | 0 | 0
Not completed — Randomized in error | 0 | 0 | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD3355 60 mg | AZD3355 120 mg | AZD3355 180 mg | AZD3355 240 mg | Placebo | Total
Number analyzed (Participants) | 134 | 125 | 136 | 126 | 140 | 661
Age Continuous [Mean (Standard Deviation); unit: years] | 47.4 (12.3) | 46.1 (13.5) | 48.0 (12.3) | 48.5 (12.1) | 48.3 (12.0) | 47.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 75 | 75 | 75 | 67 | 376
  Male | 50 | 50 | 61 | 51 | 73 | 285

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Change in GERD Symptoms Corresponding to at Least Three More Days of Not More Than Mild Symptoms on Average Per Week During Treatment (Approximately 4 Weeks) Than During Baseline (the 7 Days Before Randomisation)
Description: Symptom intensity rated by participants twice daily on a six-graded Likert scale (Did not have; Very mild; Mild; Moderate; Moderately severe; Severe) using an electronic Reflux Symptom Questionnaire diary.
  (GERD = Gastroesophageal Reflux Disease)
Time Frame: The 7 days before randomisation (baseline) and during 26-30 days of treatment
Measure: Number; unit: Participants
Arm/Group | AZD3355 60 mg | AZD3355 120 mg | AZD3355 180 mg | AZD3355 240 mg | Placebo
Number analyzed (Participants) | 134 | 125 | 136 | 126 | 140
Participants | 28 | 32 | 32 | 33 | 25

2. Secondary Outcome: Absolute Change From Baseline to Treatment Period in Percent Days With at Most Mild GERD Symptoms.
Description: Symptom intensity rated by participants twice daily on a six-graded Likert scale (Did not have; Very mild; Mild; Moderate; Moderately severe; Severe) using an electronic Reflux Symptom Questionnaire diary
  (GERD = Gastroesophageal Reflux Disease)
Time Frame: The 7 days before randomisation (baseline) and during 26-30 days of treatment
Measure: Median (Inter-Quartile Range); unit: Percent
Arm/Group | AZD3355 60 mg | AZD3355 120 mg | AZD3355 180 mg | AZD3355 240 mg | Placebo
Number analyzed (Participants) | 132 | 117 | 133 | 123 | 135
Percent | 10.7 [0 to 35.7] | 17.2 [0 to 46.4] | 11.9 [0 to 40.9] | 12.5 [0 to 47.1] | 0 [0 to 30.8]

ADVERSE EVENTS:
Description: As a consequence of the definition of the analysis set for efficacy analysis and safety analysis respectively, one patient was included in the 120 mg group for efficacy analyses and in the 60 mg group for safety analyses.
Arm/Group | AZD3355 60 mg | AZD3355 120 mg | AZD3355 180 mg | AZD3355 240 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0 | 0 | 0 | 1 | 1
Other Adverse Events (participants affected / at risk) | 13 | 12 | 16 | 20 | 9
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | AZD3355 60 mg | AZD3355 120 mg | AZD3355 180 mg | AZD3355 240 mg | Placebo
Non-Cardiac Chest Pain (General disorders) | 0/135 | 0/124 | 0/136 | 1/126 | 0/140
Metastatic Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/135 | 0/124 | 0/136 | 0/126 | 1/140
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | AZD3355 60 mg | AZD3355 120 mg | AZD3355 180 mg | AZD3355 240 mg | Placebo
Diarrhoea (Gastrointestinal disorders) | 5/135 | 7/124 | 6/136 | 10/126 | 1/140
Paraesthesia (Nervous system disorders) | 8/135 | 5/124 | 10/136 | 11/126 | 8/140

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between PI and Sponsor (AZ) or its agents that restricts the PI's right to discuss/publish trial results after the trial is completed.The PI agrees to collaborate in good faith with AZ with regards to content and formation of any publication or disclosure to be made by PI and to pay due consideration to opinions offered by AZ.